CLINICAL TRIAL: NCT04634994
Title: Novel Assessment of Synaptic Density in Progressive MS
Brief Title: Assessment of Synaptic Density in MS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, TARUN SINGHAL, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P003171
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Synaptic Density; Positron Emission Tomography; PET
MeSH Terms: conditions — Multiple Sclerosis | interventions — SynVesT-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PMS, RRMS, and Healthy Control Subjects (Experimental)
  Interventions: Drug: [F-18]SDM-8

INTERVENTIONS:
Drug: [F-18]SDM-8 — PET radiopharmaceutical. Subjects will undergo [F-18]SDM-8 PET Scanning to measure synaptic density.

SUMMARY:
The investigators propose to use the novel SV2a-PET ligand, [F-18]SDM-8 to assess synaptic density in progressive multiple sclerosis (PMS) (including primary progressive multiple sclerosis (PPMS) and secondary progressive multiple sclerosis (SPMS)), given its improved imaging characteristics and potential for large scale applicability.

The specific aims of the study are:

Aim 1: To compare the cortical and subcortical grey matter synaptic density in PMS patients, patients with relapsing-remitting MS (RRMS), and healthy subjects, using a novel [F-18] labeled synaptic density PET ligand, [F-18]SDM8, also known as [F-18]SynvesT-1.

Aim 2: To compare the relationship of synaptic density PET and standard 3T MRI measures including global and regional brain atrophy and lesion load with clinical measures of physical disability, cognitive impairment, fatigue and depression in MS patients.

Aim 3: To assess the relationship of synaptic density PET with serum neurofilament light chain (NfL) and with serum measurements of inflammatory markers, IL-1β, TNF-α, IL-6, MCP-1 (Monocyte Chemoattractant Protein-1) and MIF-1 (Macrophage Migration Inhibitory Factor-1).

DETAILED DESCRIPTION:
This is a single center, cross-sectional study of synaptic density measurement in patients with progressive MS as compared to RRMS and healthy controls.

Three groups of subjects will be recruited:

1. Subjects meeting the definition for PMS (PPMS or SPMS) by International Panel Criteria
2. Subjects meeting the definition for RRMS by the International Panel Criteria,
3. Healthy Controls

Sample Size: We plan to enroll 40 subjects including at least 10 with PMS (PPMS or SPMS), 10 with RRMS and 10 healthy controls. This is a pilot study and the sample size estimations are not based on power calculations. In order to attain our goal sample size of 30 subjects, we estimate that we may need to enroll approximately 40 subjects to account for screen failures.

Physicians at the Brigham MS Center may present the study to a subject during a regular scheduled clinic visit. If the subject is interested in the study, a copy of the consent form will be given. The subject will then be contacted by telephone prior to the screening visit appointment. At the time of the subject's screening visit, an investigator will go over the study in detail, answer any questions the subject may have regarding the study and a licensed physician investigator will obtain informed consent. In accordance with NIH guidelines, efforts will be made to attain a mix of study participants, in terms of gender and racial/ethnic representation.

Subjects may be required to come for up to 4 visits for this study.

Initial Visit:

During the first visit, subjects will be administered the screening questionnaire (if that has not already been done over telephone). Subjects will review and sign the consent form. They will be administered standardized questionnaires for cognitive testing and/or other co-morbidities.

PET Visit:

All subjects will undergo one visit for the PET scan. During the PET scan visits, all women subjects of child bearing age will undergo a stat quantitative serum hCG pregnancy test (or urine pregnancy test) and only women with a negative test will undergo the radiopharmaceutical injection.

PET imaging procedures

For PET scanning, an intravenous (IV) catheter will be inserted into the radial antecubital or other arm or hand vein for injection of tracer. Radiopharmaceutical will be injected as a bolus (approximately 5mCi for [F-18]SynVest-1 followed by 5 mL of saline).

The whole PET session will last up to 120 min.

MRI Visit:

All subjects will undergo a 3T Brain MRI during an MRI visit that may precede or follow the PET scan visit.

Pregnancy screening prior to MRI:

All women will be queried about their pregnancy status, use of contraception and last menstrual period. If they are reliably using contraception, can state the timing of their last menstrual period, and do not believe they could be pregnant, we will proceed with the MRI scan without pregnancy testing. If they cannot do this, then they will undergo a urine pregnancy test. If a woman is seeking pregnancy and not using contraception, she will undergo a urine pregnancy test.

MRI imaging procedures MRI scanning session will be performed at BWH MRI facility at 60 Fenwood Road, Boston, MA.

Several pulse sequences will be performed to image the brain. There will be no intravenous contrast used for any of the MRIs.

The MRI scan session will take approximately 1 hour.

A non-diagnostic CT scan will be performed for attenuation correction of PET transmission data at the time of initiation of scanning.

For the PET portion, as this drug is radioactive, the subject will be exposed to a small amount of radiation as a result of participation in this study. The per unit radiation dose for [F-18]SynVEst-1 is 1.4mSv/mCi_(37.8 μSv/MBq). The total amount of radiation exposure from [F-18]SynVEst-1 is 7mSv (for 5mCi injected dose). This amount of radiation is approximately 14% of the yearly amount of radiation allowed for persons who work with radiation. Additional dose from low dose CT performed for attenuation correction of PET images is estimated to be 1mSv per CT scan. Hence, the total radiation exposure from the procedure is 8mSv or approximately 16% of the yearly amount of radiation exposure allowed for persons working with radiation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the definition for MS (including PPMS, RRMS or SPMS) by International Panel (2017 McDonald) Criteria. Age and sex-matched healthy controls will also be recruited.
* Subjects willing to undergo PET and MRI imaging
* Subjects willing and able to give informed consent

Exclusion Criteria:

* Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
* Individuals with bipolar disease and schizophrenia
* Concurrent medical conditions that contraindicate study procedures.
* Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
* Claustrophobia
* Non-MRI compatible implanted devices
* Corticosteroid treatment in the past four weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PET measurements in individuals with PMS, RRMS, and healthy controls | Baseline
  To compare PET measurements including standardized uptake value (SUV) and standardized uptake value ratio (SUVR) in individuals with PMS, RRMS, and healthy controls.

SECONDARY OUTCOMES:
Correlations between PET measurements and clinical, MRI, and blood and serum measures | Baseline
  To examine correlations between PET measurements and clinical measures (e.g., Expanded Disability Status Scale, Timed 25 Foot Walk, Symbol Digit Modalities Test), MRI measures (e.g., global atrophy, regional atrophy, lesion load), and blood and serum biomarkers (e.g., nNfL).

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tourdias T, Dousset V. Neuroinflammatory imaging biomarkers: relevance to multiple sclerosis and its therapy. Neurotherapeutics. 2013 Jan;10(1):111-23. doi: 10.1007/s13311-012-0155-4. PMID 23132327
- [Background] Mendoza-Torreblanca JG, Vanoye-Carlo A, Phillips-Farfan BV, Carmona-Aparicio L, Gomez-Lira G. Synaptic vesicle protein 2A: basic facts and role in synaptic function. Eur J Neurosci. 2013 Dec;38(11):3529-39. doi: 10.1111/ejn.12360. Epub 2013 Sep 16. PMID 24102679
- [Background] Cai Z, Li S, Matuskey D, Nabulsi N, Huang Y. PET imaging of synaptic density: A new tool for investigation of neuropsychiatric diseases. Neurosci Lett. 2019 Jan 19;691:44-50. doi: 10.1016/j.neulet.2018.07.038. Epub 2018 Jul 31. PMID 30075287
- [Background] Wegner C, Esiri MM, Chance SA, Palace J, Matthews PM. Neocortical neuronal, synaptic, and glial loss in multiple sclerosis. Neurology. 2006 Sep 26;67(6):960-7. doi: 10.1212/01.wnl.0000237551.26858.39. PMID 17000961
- [Background] Mandolesi G, Grasselli G, Musumeci G, Centonze D. Cognitive deficits in experimental autoimmune encephalomyelitis: neuroinflammation and synaptic degeneration. Neurol Sci. 2010 Nov;31(Suppl 2):S255-9. doi: 10.1007/s10072-010-0369-3. PMID 20635112
- [Background] Di Filippo M, Portaccio E, Mancini A, Calabresi P. Multiple sclerosis and cognition: synaptic failure and network dysfunction. Nat Rev Neurosci. 2018 Oct;19(10):599-609. doi: 10.1038/s41583-018-0053-9. PMID 30158590
- [Background] Friese MA. Widespread synaptic loss in multiple sclerosis. Brain. 2016 Jan;139(Pt 1):2-4. doi: 10.1093/brain/awv349. No abstract available. PMID 26747852
- [Background] Peterson JW, Bo L, Mork S, Chang A, Trapp BD. Transected neurites, apoptotic neurons, and reduced inflammation in cortical multiple sclerosis lesions. Ann Neurol. 2001 Sep;50(3):389-400. doi: 10.1002/ana.1123. PMID 11558796
- [Background] Weiner HL. The challenge of multiple sclerosis: how do we cure a chronic heterogeneous disease? Ann Neurol. 2009 Mar;65(3):239-48. doi: 10.1002/ana.21640. PMID 19334069